CLINICAL TRIAL: NCT06119516
Title: Transpulmonary Pressure - Guided Mechanical Ventilation in Morbidly Obese ARDS Patients: a Feasibility Study.
Acronym: TGV-MOA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APHP220824; 2023-A01044-41 (Other: Agence nationale de sécurité du médicament et des produits de santé); PHRC21-0254 (Other Grant/Funding Number: French Ministry of health); DR-2023-130 (Other: Commission Nationale de l'Informatique et des Libertés)
Record Dates: First submitted 2023-10-12; First posted 2023-11-07 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: ARDS, Human; Obesity, Morbid
Keywords: ARDS, Human; Obesity, morbid; Mechanical Ventilation; Transpulmonary pressure
MeSH Terms: conditions — Respiratory Distress Syndrome; Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Esophageal pressure-guided strategy, (Experimental): The second generation esogastric multifunction Nutrivent catheter (SIDAM, Mirandola, Italy) will be used to monitor esophageal and gastric pressures during several days. Ventilator settings will be adjusted to the evaluated esophageal pressure-guided strategy, aiming to obtain a slightly positive transpulmonary pressure at the end of expiration.
  Interventions: Other: Esophageal pressure-guided strategy,

INTERVENTIONS:
Other: Esophageal pressure-guided strategy, — A catheter-balloon system will be positioned and calibrated in all included patients. The second generation esogastric multifunction Nutrivent catheter (SIDAM, Mirandola, Italy) will be used. It allows both enteral nutrition of the patients and monitoring of esophageal and gastric pressures during several days. A connection line will be inserted between the catheter (either esophageal or gastric balloon port) and the auxiliary pressure port of the mechanical ventilator (General Electric, R860, available in each center). Numeric recording of the respiratory signals will be achieved via the OhmedaCom Research Tool software, helping for centralization of the analyses, therefore ensuring reproducibility of the results.

SUMMARY:
The goal of this clinical trial is to test a personalized intervention aiming to optimize the mechanical ventilator settings in morbidly obese patients suffering from moderate to severe Acute Respiratory Distress Syndrome (ARDS). The intervention consists of personalized measurements and calculations of the different pressures inside the thorax. The main question to answer is:

• Will the evaluated esophageal pressure-guided strategy lead to different mechanical ventilator settings than suggested by a strategy largely used in ARDS patients in France?

A specific nasogastric probe permitting to measure esophageal pressure will monitor participants. Esophageal pressure will act as an indicator of the pleural pressure. Other respiratory signals displayed by the mechanical ventilators will also be acquired.

Further, ventilator settings will be adjusted to the evaluated esophageal pressure-guided strategy, with possible benefit of this personalized approach.

DETAILED DESCRIPTION:
The goal of this clinical trial is to test a personalized intervention aiming to optimize the mechanical ventilator settings in morbidly obese patients suffering from moderate to severe Acute Respiratory Distress Syndrome (ARDS). Mechanical ventilation is the cornerstone of the ARDS symptomatic treatment. Individualization of mechanical ventilator settings could improve prognosis mainly by preventing or decreasing accumulation of fluid in the lung and hemodynamic impairment. It is likely that class III obesity ARDS patients (defined by body mass index (BMI) > 40 kg/m2), could benefit from a highly personalized approach, based on esophageal pressure monitoring. These patients have significantly higher esophageal pressures, acting as an indicator of pleural pressure, than the general ARDS population, while these patients have rather normal mechanical characteristics of the chest wall. Such features could suggest innovative mechanical ventilator settings, by integrating esophageal pressures values, aiming to obtain a slightly positive transpulmonary pressure at the end of expiration.

The intervention consists of personalized measurements and calculations of the different pressures, including the esophageal one, inside the thorax.

The main question to answer is:

• Will the evaluated esophageal pressure-guided strategy lead to different mechanical ventilator settings, mainly the positive end-expiratory pressure (PEEP) setting, than suggested by a PEEP-strategy largely used in ARDS patients in France?

A specific nasogastric probe permitting to measure esophageal pressure will monitor participants. The second generation esogastric multifunction Nutrivent catheter (SIDAM, Mirandola, Italy) will be used. It allows both enteral nutrition of the patients and monitoring of esophageal and gastric pressures during several days. Esophageal pressure will act as an indicator of the pleural pressure. Other respiratory signals displayed by the mechanical ventilators will also be acquired, permitting to calculate the trans-pulmonary pressures.

Further, ventilator settings will be adjusted to the evaluated esophageal pressure-guided strategy, with possible benefits of this personalized approach. The main benefits for the research participants will be the application of highly personalized mechanical ventilator settings, aiming mainly to select the best PEEP setting with the goal of optimization of opening the lung while avoiding the respiratory and hemodynamic consequences of excessive lung inflation. Monitoring of the end-inspiratory transpulmonary pressures will help to prevent excessive lung inflation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (aged 18 years or older)
* Class III morbid obesity (BMI > 40 kg/m2)
* Moderate or severe ARDS criteria (according to the Berlin definition)
* Less than 72 hours between fulfilling moderate or severe ARDS criteria and inclusion
* Tracheal intubation and invasive mechanical ventilation
* Informed consent (patient, next of kin), with possibility of an emergency procedure with deferred consent
* Covid-19 and non-Covid-19 patients

Exclusion Criteria:

* Contra-indication to nasogastric tube (uncontrolled coagulopathy, severe thrombocytopenia, nasal trauma, esophageal varices)
* Order to limit life-sustaining therapy
* ExtraCorporal Membrane Oxygenation (ECMO) in use
* Invasive mechanical ventilation > 96 hours
* Elevated intracranial pressure
* Active air-leak: pneumothorax, pneumomediastinum
* Pregnancy or breast feeding
* Patient on state medical aid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-04-04 (Actual); Primary Completion 2026-04-04 (Estimated); Study Completion 2026-07-04 (Estimated)

PRIMARY OUTCOMES:
The absolute value of the difference between the PEEP levels determined by esophageal pressure-guided strategy and by the PEEP level indicated by the maximal recruitment arm of the ExPress trial | during the first 24 hours after inclusion
  To demonstrate that the evaluated esophageal pressure-guided strategy leads to significantly and clinically different mechanical ventilator settings (mainly PEEP setting) than the reference strategy.

SECONDARY OUTCOMES:
The ratio between the arterial partial pressure of oxygen (PaO2) on the inspired fraction of oxygenFiO2): PaO2/FiO2 ratio | during the intervention
  To assess the efficacy of the esophageal pressure-guided strategy.
The mortality rate of included patients. | Mortality rate will be determined at end of ICU stay, at Day 28 and at Day 90.
  To assess the efficacy and safety of the esophageal pressure-guided strategy.
Number of days alive and free for invasive mechanical ventilation | The numbers of days alive and free for invasive mechanical ventilationwill be determined at Day-28 and Day-90
  To assess the efficacy of the esophageal pressure-guided strategy.
Occurrence of pneumothorax | during the intervention
  To assess the safety of the esophageal pressure-guided strategy.
Occurence of severe hemodynamic compromise defined by the need of vasoactive treatment | during the intervention
  To assess the safety of the esophageal pressure-guided strategy.
Percentage of included patients with inability to insert the Nutrivent catheter | during the first 24 hours after inclusion
  To assess the feasibility of the esophageal pressure-guided strategy.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc MD Diehl, PhD, Study Chair — AP-HP, Hôpital Européen Georges Pompidou, Paris
Locations (5):
- France (5):
  - CHU Angers, Angers
  - Hôpital Bicêtre, AP-HP, Le Kremlin-Bicêtre
  - Hôpital de la Croix-Rousse, HCL, Lyon
  - AP-HP, Hôpital Européen Georges Pompidou, Paris
  - CHU la Milétrie, Poitiers

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie results in publication could be shared. IPD detailed in the protocol of a planned metaanalysis could be shared
Supporting Information: Study Protocol, ICF
Time Frame: Two years after the last publication
Access Criteria: Data sharing must be accepted by the sponsor and the PI based on a scientific project and scientific involvement of the PI team. Collaboration will be fostered. The founder could be involved in the decision.
  Teams wishing obtain IPD must meet the sponsor and IP team to present scientifics (and commercial) purpose, IPD needed, format of data transmission, and timeframe. Technical feasibility and financial support will be discussed before mandatory contractualization.
  Processing of shared data must comply with European General Data Protection Regulation (GDPR).

REFERENCES:
- [Background] Diehl JL, Talmor D. When could airway plateau pressure above 30 cmH2O be acceptable in ARDS patients? Intensive Care Med. 2021 Sep;47(9):1028-1031. doi: 10.1007/s00134-021-06472-5. Epub 2021 Jul 8. No abstract available. PMID 34236478
- [Result] Coudroy R, Vimpere D, Aissaoui N, Younan R, Bailleul C, Couteau-Chardon A, Lancelot A, Guerot E, Chen L, Brochard L, Diehl JL. Prevalence of Complete Airway Closure According to Body Mass Index in Acute Respiratory Distress Syndrome. Anesthesiology. 2020 Oct 1;133(4):867-878. doi: 10.1097/ALN.0000000000003444. PMID 32701573
- [Result] Florio G, Ferrari M, Bittner EA, De Santis Santiago R, Pirrone M, Fumagalli J, Teggia Droghi M, Mietto C, Pinciroli R, Berg S, Bagchi A, Shelton K, Kuo A, Lai Y, Sonny A, Lai P, Hibbert K, Kwo J, Pino RM, Wiener-Kronish J, Amato MBP, Arora P, Kacmarek RM, Berra L; investigators of the lung rescue team. A lung rescue team improves survival in obesity with acute respiratory distress syndrome. Crit Care. 2020 Jan 15;24(1):4. doi: 10.1186/s13054-019-2709-x. PMID 31937345
- [Result] Rowley DD, Arrington SR, Enfield KB, Lamb KD, Kadl A, Davis JP, Theodore DJ. Transpulmonary Pressure-Guided Lung-Protective Ventilation Improves Pulmonary Mechanics and Oxygenation Among Obese Subjects on Mechanical Ventilation. Respir Care. 2021 Jul;66(7):1049-1058. doi: 10.4187/respcare.08686. Epub 2021 Apr 20. PMID 33879565
- [Result] Sarge T, Baedorf-Kassis E, Banner-Goodspeed V, Novack V, Loring SH, Gong MN, Cook D, Talmor D, Beitler JR; EPVent-2 Study Group. Effect of Esophageal Pressure-guided Positive End-Expiratory Pressure on Survival from Acute Respiratory Distress Syndrome: A Risk-based and Mechanistic Reanalysis of the EPVent-2 Trial. Am J Respir Crit Care Med. 2021 Nov 15;204(10):1153-1163. doi: 10.1164/rccm.202009-3539OC. PMID 34464237